CLINICAL TRIAL: NCT07183319
Title: Circulating Tumor DNA Response Adapted Treatment De-escalation Metastatic Urothelial Carcinoma (CT-READ)
Brief Title: Circulating Tumor DNA Response In Urothelial Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-CT-READ
Record Dates: First submitted 2025-09-02; First posted 2025-09-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Urothelial Carcinoma
Keywords: Metastatic; ctDNA; Pembrolizumab; De-escalation therapy
MeSH Terms: conditions — Carcinoma, Transitional Cell; Neoplasm Metastasis | interventions — pembrolizumab; enfortumab vedotin

STUDY DESIGN:
Intervention Model Description: This study is a single-arm, open-label pilot trial evaluating de-escalation of therapy in patients with reduction in ctDNA following 1L Pembrolizumab & Enfortumab Vedotin (PEV) for Metastatic Urothelial Carcinoma (mUC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab & Enfortumab Vedotin (PEV) (Experimental): Patients with metastatic urothelial carcinoma (mUC) will initiate first-line (1L) PEV therapy as the standard of care. At 24 weeks, radiographic imaging will be performed to evaluate disease status. Patients who exhibit either stable disease or ongoing radiographic response, accompanied by a ≥50% reduction in circulating tumor DNA (ctDNA) levels, will transition to pembrolizumab monotherapy as part of a treatment de-escalation strategy. Pembrolizumab will be continued until the occurrence of disease progression or unacceptable toxicity. In the event of progression or intolerance, patients will be re-challenged with first-line PEV therapy and continue treatment until completion of the study-defined treatment period.
  Interventions: Drug: Pembrolizumab & Enfortumab Vedotin (PEV); Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab & Enfortumab Vedotin (PEV) — Patients in the study will receive 1L PEV with 1.25 mg/kg of EV on day 1 and day 8 every 21 days, and 200 mg of pembrolizumab every 21 days.
  Other Names: PADCEV
Drug: Pembrolizumab — Patients will receive 400 mg of pembrolizumab every 42 days. During the de-escalation period from PEV.
  Other Names: KEYTRUDA
Drug: Pembrolizumab & Enfortumab Vedotin (PEV) — If patients experience radiographic progression on pembrolizumab monotherapy, they will undergo rechallenge with PEV.
  Other Names: PADCEV

SUMMARY:
The purpose of this clinical trial is to evaluate the effectiveness of pembrolizumab monotherapy following 24 weeks of frontline pembrolizumab & Enfortumab Vedotin (PEV) in patients with metastatic urothelial cancer (mUC).

DETAILED DESCRIPTION:
This study aims to evaluate the de-escalation of therapy in patients with metastatic urothelial carcinoma (mUC). Patients will begin treatment with first-line (1L) (PEV) per standard of care. After 24 weeks, patients will be assessed for disease progression. Those who demonstrate stable disease or ongoing disease radiographic response and a ≥50% reduction in circulating tumor DNA (ctDNA) levels will enter the de-escalation phase. This phase consists of transitioning from PEV to pembrolizumab monotherapy. If, during the de-escalation period, patients exhibit disease progression or increased toxicity, they will be rechallenged with PEV.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically documented unresectable, locally advanced, or metastatic urothelial carcinoma.
* Measurable disease according to the New Response Evaluation Criteria in Solid Tumors (RECIST v1.1)38

  a. Participants with prior definitive radiation therapy must have measurable disease per RECIST v1.1 that is outside the radiation field or has demonstrated unequivocal progression since completion of radiation therapy.
* Must be considered eligible to receive cisplatin- or carboplatin-containing chemotherapy, in the investigator's judgment.
* Archival tumor tissue comprising muscle-invasive urothelial carcinoma, or a biopsy of metastatic urothelial carcinoma must be available for tumor-informed ctDNA analysis.
* Meets Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1, or 2.
* Adequate hematologic and organ function (Hb ≥ 8.0 g/dL; ANC ≥ 1.5x109 cells/L; CrCl ~30 mL/min; total bilirubin ≤ 1.5 mg/dL; ALT and AST within normal limits).

Exclusion Criteria:

* Previously received enfortumab, vedotin, or other monomethyl auristatin E (MMAE)-based ADCs.
* Received prior treatment with a programmed cell death ligand-1 (PD-(L)-1) inhibitor for any malignancy, including earlier stage UC, defined as a PD-1 inhibitor or PD-L1 inhibitor within 12 months.
* Has received anti-cancer treatment with chemotherapy, biologics, or investigational agents not otherwise prohibited by exclusion criterion 1-3 that is not completed within 28 days prior to cycle 1 day 1.
* Has uncontrolled diabetes or ≥ grade III peripheral neuropathy.
* Patient's estimated life expectancy is less than 12 weeks.
* Has untreated central nervous system metastases.
* Experiences ongoing clinically significant toxicity associated with prior treatment that has not resolved to ≤ Grade 1 or returned to baseline.
* Is currently receiving systemic antimicrobial treatment for active infection (viral, bacterial, or fungal). Routine antimicrobial prophylaxis is permitted.
* Has known active hepatitis B, active hepatitis C, or human immunodeficiency virus (HIV) infection.
* Has history of another invasive malignancy requiring treatment within 3 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy (excluding localized prostate cancer or basal cell carcinoma of skin or squamous cell carcinoma of the skin).
* Has documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association (NYHA) Class IV within 6 months.
* Received radiotherapy within 2 weeks.
* Received major surgery (defined as requiring general anesthesia and >24-hour inpatient hospitalization) within 2 weeks.
* Known severe (≥ Grade 3) hypersensitivity to any EV excipient contained in the drug formulation of EV.
* Has active keratitis or corneal ulcerations.
* Has a history of autoimmune disease that has required systemic immunosupressive treatment in the past 2 years, or uncontrolled autoimmune disease.
* Participants must not have received prior systemic therapy for locally advanced or metastatic urothelial carcinoma with the following exceptions:

  * Participants that received neoadjuvant chemotherapy with recurrence >12 months from completion of therapy are permitted.
  * Participants that received adjuvant chemotherapy or ICPIs therapy following cystectomy with recurrence >12 months from completion of therapy are permitted.
* Has a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.
* Has received prior allogeneic stem cell or solid organ transplant.
* Received a live attenuated vaccine within 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
3 months of progression-free survival (PFS) while on Pembrolizumab Monotherapy. | 3 months
  Number of patients who achieve PFS at the 3-month mark on pembrolizumab monotherapy. These patients will undergo radiographic assessments to evaluate progression-free survival (PFS).
6 months of PFS while on Pembrolizumab Monotherapy | 6 months
  Number of patients in the de-escalation phase who have reached 6-month PFS while on pembrolizumab monotherapy.

SECONDARY OUTCOMES:
Treatment Related Adverse Events (TRAEs) while on Pembrolizumab Monotherapy. | 1 year
  Number of patients who experience treatment-related adverse events (TRAEs) while in the de-escalation phase treated with pembrolizumab monotherapy following 1L PEV. Any adverse events (AEs) or TRAEs that do occur will be assessed and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Pain Assessment In Patients While On Pembrolizumab Monotherapy. | 1 year
  The Brief Pain Inventory (BPI) questionnaire will be administered to assess participants' perceived pain levels. Pain intensity will be rated on a Likert scale ranging from 0, indicating no pain, to 10, representing the most severe and unimaginable pain.
Changes In Peripheral Neuropathy While on Pembrolizumab Monotherapy | 1 year
  The Functional Assessment of Cancer Therapy-Neurotoxicity 12 (FACT-NTX-12) will be administered every 12 weeks to evaluate peripheral neuropathy. This tool measures quality of life in relation to neuropathy symptoms, vibration perception threshold, and extension strength testing. Responses are rated on a 5-point Likert scale, ranging from 0 ("not at all") to 4 ("very much").
Health Assessment In Patients While On Pembrolizumab Monotherapy | 1 year
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) will be administered to assess participants' quality of life, including physical, emotional, and social functioning, as well as cancer-related symptoms. Responses are measured on a Likert scale from 1 ("not at all") to 4 ("very much").

CONTACTS AND LOCATIONS:
Overall Officials: Adanma Ayanambakkam, MD, Principal Investigator — University of Oklahoma
Locations (1):
- OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No